CLINICAL TRIAL: NCT06752382
Title: Sintilimab Combined With Bevacizumab and Induction Chemotherapy in the Treatment of High Risk Advanced Nasopharyngeal Carcinoma Prospective, Single-arm, Multicenter Phase II Clinical Study
Brief Title: Sintilimab Combined With Bevacizumab and TP Chemotherapy in the Treatment of High Risk Locally-advanced NPC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Jiang Feng, Director, department of head and neck radiotherapy, Principal Investigator, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2024-363
Record Dates: First submitted 2024-12-11; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Locally Advanced Nasopharyngeal Carcinoma
Keywords: PD-1; Bevacizumab; TP Chemotherapy
MeSH Terms: interventions — Drugs, Investigational

STUDY DESIGN:
Intervention Model Description: Eligible enrolled patients will receive 3 cycles of induction therapy: sintilimab, bevacizumab, and TP regimen chemotherapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental (Experimental): Eligible enrolled patients will receive 3 cycles of induction Guided treatment and concurrent chemoradiotherapy. Then all patients received 2 cycles of concurrent chemoradiotherapy cisplatin 100mg/m2 with Intensity modulated radiotherapy for 70Gy/33Fr.Then patients received sintilimab 200mg IV every three weeks with no more than 8 cycles.
  Interventions: Drug: Experimental drug

INTERVENTIONS:
Drug: Experimental drug — Induction therapy was sintilimab 200mg IV d1, bevacizumab 7.5mg/kg IV d1, albumin-bound paclitaxel 260mg/m2 IV d1 and cisplatin 80mg/m2 IV d1, once every 3 weeks, a total of 3 cycles.
  Other Names: sintilimab ,bevacizumab and TP chemotherapy

SUMMARY:
Nearly half of the world's nasopharyngeal cancer occurs in China, among which the highest incidence in Guangdong and Guangxi, so the nickname "Guangdong tumor". Due to the hidden position of the nasopharynx, 70% to 80% of patients are found in the middle and late stages. Immunotherapy plays a significant role in nasopharyngeal carcinoma. Professor Ma Jun of Sun Yat-sen University reported a phase 3 clinical study at ASCO meeting in 2023, which compared the efficacy of Sintilimab combined with GP chemotherapy versus GP chemotherapy alone in locally advanced nasopharyngeal carcinoma, and the results showed that EFS in the immune group decreased by 41% in 3 years. The risk of local recurrence-free survival and distant metastasis was reduced by 48% and 43%, respectively. However, a subgroup analysis of the study found that low-risk patients benefited more, while N2-N3 patients benefited only HR There is 0.78, new treatment options need to be explored in clinic. Therefore, the investigators plan to initiate a prospective study to evaluate the efficacy and safety of Sintilimab Combined With Bevacizumab and TP Chemotherapy for high-risk locally advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, multicenter, Phase II clinical study. This study was planned to include patients with histologically confirmed non-keratinized stage TanyN2-3M0 nasopharyngeal carcinoma (AJCC Version 8). Eligible enrolled patients will receive 3 cycles of induction therapy: sintilimab, bevacizumab, and TP regimen chemotherapy. After induction therapy, all patients received radical concurrent chemoradiotherapy and maintenance treatment with sintilimab.The primary endpoint is radiographic complete response rate after induction therapy.The secondary endpoint are two years PFS rate and safety which is the incidence and severity of AE evaluated according to the NCI CTCAE (version 5.0) classification of the severity of adverse events, and the correlation with the study drugs was analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Signed a written informed consent form (ICF) voluntarily.
2. Male or female, aged from 18 to 75 years.
3. Histologically newly diagnosed patients with differentiated or undifferentiated non-keratinous carcinoma (according to World Health Organization [WHO] histological types).
4. Patients with tumor stage TanyN2-3M0 (according to AJCC Edition 8).
5. ECOG score 0-1.
6. Adequate bone marrow/liver and kidney function/heart and lung and other physiological function reserves, expected to successfully complete chemoradiotherapy and immunotherapy.

Exclusion Criteria:

1. subjects with pathologically diagnosed adenocarcinoma or sarcoma of the nasopharynx.
2. subject has other malignancy within 3 years prior to first dose except nasopharyngeal carcinoma. Subjects with other malignancies that have been cured by local therapy, such as basal or cutaneous squamous cell carcinoma, superficial bladder cancer, cervical or breast carcinoma in situ, are excluded.
3. Participated in treatment with an investigational drug or used an investigational device within 4 weeks prior to the first dose.
4. active or previous definite inflammatory bowel disease (e.g., Crohn 's disease or ulcerative colitis) disease.
5. History of immunodeficiency; positive HIV antibody test; current chronic use of systemic corticosteroids or other immunosuppressive agents; local, ocular, intra-articular, intranasal, and inhaled corticosteroids are allowed.
6. Patients who are pregnant or nursing (for women of childbearing age, pregnancy testing should be considered and the use of effective contraception during treatment should be emphasized).
7. Subjects with known active pulmonary tuberculosis (TB) and suspected active TB require clinical examination to rule out; known active syphilis infection.
8. known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation; 9. history of pneumonitis/interstitial lung disease requiring systemic corticosteroids or current pneumonitis.
9. serious infections within 4 weeks prior to the first dose, including but not limited to comorbidities requiring hospitalization, sepsis, or serious pneumonia; active infections (excluding antiviral therapy for hepatitis B or C) that have received systemic anti-infective therapy within 2 weeks prior to the first dose.
10. Subjects with untreated active hepatitis B (HBsAg positive and HBV-DNA more than 1000 copies/ml [200 IU/ml] or above the lower limit of detection) and anti-hepatitis B virus treatment during study treatment are required for subjects with hepatitis B; subjects with active hepatitis C (HCV antibody positive and HCV-RNA level above the lower limit of detection).
11. any of the following cardiovascular and cerebrovascular diseases: a) myocardial infarction, unstable angina pectoris, cerebrovascular accident, transient ischemic attack, acute or persistent myocardial ischemia, symptomatic heart failure (Grade 2 and above according to the New York Heart Association functional classification), or any arterial thromboembolic event within 6 months before the first dose; b) history of venous thromboembolic events (NCI CTCAE 5.0 version 3 and above), pulmonary embolism, or other serious thromboembolism within 3 months before the first dose; c) presence of serious arrhythmia requiring long-term drug intervention; patients with asymptomatic atrial fibrillation with stable ventricular rate are allowed; d) presence of aortic aneurysm, aortic dissecting aneurysm, internal carotid artery stenosis and other major vascular diseases that may be life-threatening or require surgery within 6 months; e) previous history of myocarditis or cardiomyopathy.
12. Known hypersensitivity to any component of any study drug; known history of serious hypersensitivity to other monoclonal antibodies.

13 known history of mental illness, drug abuse, alcoholism, or drug abuse; 15. pregnant or lactating women. 16. Any previous or current illness, treatment, or laboratory abnormality that may confound the results of the study, affect the subject 's full participation in the study, or that participation may not be in the subject' s best interest.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
radiographic complete response rate | At the end of Cycle 3 (each cycle is 21 days)
  CR rate was evaluated according to recist 1.1 criteria

SECONDARY OUTCOMES:
progression-free survival | 2 years
  The time from the time the patient receives treatment to the time the disease progresses or death (whatever the cause)
AE | 2 years
  The incidence and severity of acute effects were evaluated according to the NCI CTCAE (version 5.0) classification of the severity of adverse events, and the correlation with the study drugs was analyzed. Safety and tolerability of changes in vital signs, physical examination, and laboratory tests during the study were evaluated according to the severity of adverse events (AE) according to NCI CTCAE (version 5.0).

CONTACTS AND LOCATIONS:
Overall Officials: feng jiang, PhD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No